CLINICAL TRIAL: NCT04644250
Title: Phase II of Toripalimab Chemoradiotherapy in Neoadjuvant Treatment of Locally Advanced Esophageal Squamous Cell Carcinoma: A Single-center、Open Lable、Single-arm Exploratory Clinical Research
Brief Title: Combination of Toripalimab and Neoadjuvant Chemoradiotherapy for Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wei Ren (Other)
Responsible Party: Sponsor-Investigator, Wei Ren, clinical professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLYY-EC-NAD-01
Record Dates: First submitted 2020-11-16; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Locally advanced esophageal squamous cell carcinoma; Neoadjuvant chemoradiotherapy; Radical resection; Toripalimab
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — toripalimab; Carboplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm1 (Experimental): Arm1:preoperative Toripalimab with chemoradiotherapy group Participants will receive carboplatin (AUC=2) VD 30min and paclitaxel liposome (50mg/m²) CIV 24h on day 3,10,17,24,31. And radiotherapy will start from day 1 to 31 of chemotherapy. A total of 41.4 Gy, 23 fractions of 1.8 Gy. Participants will also receive Toripalimab(240mg) VD 30 min on days 3, 24 and 45. After the above neoadjuvant therapy is over, the short-term efficacy evaluation will be performed first, and then a scheduled radical radical resection will be performed from days 59 to 73.
  Interventions: Drug: Toripalimab; Drug: Paclitaxel liposome/Carboplatin; Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Toripalimab — Participants will also receive Toripalimab(240mg) VD 30 min on days 3, 24 and 45，3 cycles in total.
  Other Names: JS-001
Drug: Paclitaxel liposome/Carboplatin — Participants will receive carboplatin (AUC=2) VD 30min and paclitaxel liposome (50mg/m²) CIV 24h on day 3,10,17,24,31, 5cycles in total.
  Other Names: PCb
Radiation: Intensity-modulated radiotherapy — A total of 41.4 Gy, 23 fractions of 1.8 Gy on Day 1 to 31.
  Other Names: IMRT

SUMMARY:
Radical resection is thought to be the mainstay of esophageal cancer treatment. Neoadjuvant chemoradiotherapy (CRT) followed by surgery has become the standard treatment option for locally advanced esophageal squamous cell cancer (ESCC). However, only 20% to 40% of patients can achieve pathologic complete response (pCR) after neoadjuvant CRT with favorable prognosis and about 10% of patients have disease progression after chemoradiotherapy. How to improve the the efficacy of neoadjuvant therapy is an important clinical problem to be solved.

Immunotherapy targeting the programmed cell death receptor-1（PD-1） /programmed cell death-Ligand 1(PD-L1) checkpoints has demonstrated promising activity in ESCC. In Keynote181 study, for patients with metastatic esophageal squamous cell carcinoma, regardless of PD-L1 expression, pembrolizumab significantly improved overall survival compared with chemotherapy. However, the efficacy and safety of immunotherapy therapy in surgery-based multidisciplinary treatment of local advanced esophageal cancer still need a lot of clinical studies to further confirm.

This study aims to investigate the safety and efficacy of Toripalimab combined with radiotherapy and chemotherapy in neoadjuvant treatment of locally advanced esophageal squamous cell carcinoma

DETAILED DESCRIPTION:
This study was designed as an open-lable, single-arm, single-center,exploratory clinical study. Toripalimab combination of chemoradiotherapy as neoadjuvant therapy. Participants will receive carboplatin (AUC=2) and paclitaxel liposome (50mg/m²) on day 3,10,17,24,31. And radiotherapy Intensity-modulated radiation therapy（IMRT）will start from day 1 to 31 of chemotherapy. A total of 41.4 Gy, 23 fractions of 1.8 Gy. Participants will also receive Toripalimab (240mg) on days 3, 24and 45. After the neoadjuvant treatment is over, the short-term efficacy evaluation will be performed first, and then a radical resection will be scheduled on Day 59 to 73. This study include 2 phases: 14 cases were enrolled in the first stage and 18 cases were enrolled in the second stage.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years old of either gender
2. A histopathological diagnosis of resectable thoracic esophageal squamous cell carcinoma(The midpoint of the upper and lower margins of the primary tumor is ≥25cm from the incisor)
3. There is no distant metastasis and the esophageal tumor can be resected or potentially resectable after the expert consultation of thoracic surgery. The clinical stage is cT3-4aN0-2M0, patients with stage Ⅱ, Ⅲ, and IVA (AJCC 8th edition cTNM staging);
4. ECOG PS score of 0-1;
5. Patients who are anti-tumor treatment-naive;
6. Estimated life expectancy >6 months
7. Baseline the function of important organs meets the following requirements: a. white blood cell count (WBC) ≥ 3×109/L, absolute neutrophil count (ANC) ≥ 1.5×109/L，;Baseline organ function meets: ①WBC≥3×109/L, ANC≥1.5×109/L, PLT≥100×109/L, Hb≥90g/L; ②Liver function: TBIL≤2ULN, Aspartate aminotransferase（AST） ≤2.5ULN, ALT≤2.5ULN ③renal function: cCr≥60 ml/min, Cr≤1.5 ULN; ④heart function: no heart disease or coronary heart disease, the patient's heart function is 1-2 grade;
8. The blood pressure of hypertensive patients should be controlled within the normal range with antihypertensive drugs;
9. The fasting blood-glucose of diabetic patients should be controlled at ≤8mmol/L through hypoglycemic drugs;
10. No other serious diseases that conflict with this plan (such as autoimmune diseases, immunodeficiency, organ transplantation, or other diseases that require continuous hormone therapy);
11. No history of other malignant tumors;
12. The patient agrees to participate in this clinical study and signs the "Informed Consent". Ability to understand the study and sign informed consent.

Exclusion Criteria:

1. Patients who have been treated previously with anti-tumor therapy (including chemotherapy, radiotherapy, surgery, immunotherapy, etc.);
2. Patients with other malignant tumors (non-malignant black skin tumors, cervical cancer in situ, except for cured prostate cancer);
3. Patients who have been or expected to have a significant risk of esophageal perforation, fistula, and major bleeding;
4. Patients who have active autoimmune diseases or patients who are undergoing treatment of autoimmune diseases (Prior therapy with immunosuppressant, the dose of immunosuppressant used ≥10mg/day, oral prednisone for more than 2 weeks);.
5. Uncontrolled clinically significant cardiovascular and cerebrovascular diseases , including but not limited to severe acute myocardial infarction, unstable or severe angina pectoris, coronary artery bypass surgery, congestive heart failure, ventricular arrhythmia requiring medical intervention within 6 months before enrollment 、Left ventricular ejection fraction <50%, or other patients who are not expected to tolerate chemotherapy and radiotherapy;Cardiac clinical symptoms or diseases that are not well controlled, such as: a. Heart Failure（New York Heart Association）> Class Ⅱ, b. unstable angina, c. myocardial infarction within 1 year; d. Clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention.
6. Patients who were severe allergic constitution;;
7. Patients who were pregnant or lactating women;
8. Patients who have severe mental disorders;
9. Patients who have peripheral nerve disease with common terminology criteria (CTC）grade ≥3;
10. Abnormal blood coagulation function including PT>16s, activated partial thromboplastin time（APTT）>53s, Thrombin time（TT）>21s, Fib<1.5g/L, bleeding tendency or receiving thrombolytic or anticoagulant therapy;
11. Patients who hsve severe pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, severely impaired lung function, etc past or present., or active tuberculosis within 1 year;
12. Patients who have active hepatitis B or C;
13. Patients who did not meet the enrollment conditions xia researchers evaluated.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate | Three working days after surgery
  Pathologic complete response was defined as pT0N0M0（clinical stage). The rate of pathologic complete response rate after neoadjuvant chemoradiotherapy.

SECONDARY OUTCOMES:
Incidence of Treatment-related Adverse Events as Assessed by CTCAE v4.0 | From the enrollment to the date of surgery
  The neoadjuvant treatment-related adverse events
2-year overall survival | From date of randomization until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 24 months
  The 2-year overall survival of the whole group
2-year disease-free survival | From date of surgery until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 24 months.
  The 2-year disease-free survival of the whole group
Major Pathological Response (MPR) rate | From date of surgery to 14 days later
  MPR is defined as 10% or fewer viable cancer cells in the hematoxylin and eosin (H&E)-stained slides from the resected tumor following neoadjuvant treatment.
Objective Response Rate (ORR) | At the end of Cycle 2 (each cycle is 21 days)
  Objective response rate is defined as the rate of patients with at least a 30% decrease in the sum of the longest diameter of target lesions, which include complete response (CR) or partial response (PR).
R0 resection rate | Three working days after surgery
  The R0 resection rate of esophagectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No